CLINICAL TRIAL: NCT01439074
Title: An Open, Randomized, Comparative, Multi-centre Investigation Evaluating the Efficacy and Tolerance of Mepilex Ag Versus Silver Sulfadiazine in the Treatment of Deep Partial Thickness Burn Injuries.
Brief Title: Mepilex Ag Versus Silver Sulfadiazine in Children and Adults With Burn Injuries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMA 418
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2013-12

CONDITIONS: Burn Injuries
Keywords: Burn injuries; Mepilex Ag; SSD Ag; Partial thickness
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepilex Ag (Active Comparator): Mepilex Ag consists of a Safetac(R) soft silicone wound contact layer, a grey absorbent polyurethane foam pad containing a silver compound, activated carbon, and a vapour permeable waterproof film.
  Interventions: Device: Mepilex Ag
- Silver Sulphadiazine Ag cream (Active Comparator): SSD Ag cream is white cream, 1% SSD Ag, 40g/tube This cream is indicated for prevent and treat secondary wound infection of small area, mild burn/scald.
  Interventions: Drug: Silver Sulphadiazine Ag cream

INTERVENTIONS:
Device: Mepilex Ag — Dressing
  Other Names: Absorbent foam silver dressing
  Arms: Mepilex Ag
Drug: Silver Sulphadiazine Ag cream — A cream used on burnt areas.
  Other Names: SSD Ag cream, 1% SSD Ag, 40g/tube
  Arms: Silver Sulphadiazine Ag cream

SUMMARY:
The purpose is to compare time to healing using absorbent foam silver dressing (Mepilex Ag) compared to a silver sulfadiazine (SSD) 1% cream in the treatment of partial thickness burn injuries.284 in-patients in 8-12 centres in China will be evaluated. Treatment period will be up to 4 weeks with either Mepilex Ag or SSD.

DETAILED DESCRIPTION:
Subjects enrolled in this investigation were in-patients at eleven centers in China. To be included, subjects had to have deep partial-thickness burn injuries. The subjects were consecutively allocated to a subject code providing they fulfilled all inclusion criteria and none of the exclusion criteria and had signed a written informed consent form. Two evaluators independent of each other made the judgment regarding depth of the burn before enrolling a subject. The subjects were randomized to either receive Mepilex Ag or SSD.

Treatment period were up to four weeks with either SSD or Mepilex Ag. Changes of the investigation products were performed according to a standardized schedule, unless the wound healed before.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a deep partial-thickness burn injury covering 2.5%-25% TBSA (3rd degree areas not to exceed 10% TBSA)
* Burn of thermal origin
* Both gender with an age ≥5 years and ≤65 years at ICF
* Understood and signed informed consent
* Subjects who are younger than the legal consenting age must have a legally authorized representative

One study burn should be chosen which fulfil the following criteria;

1. isolated burn area (not head and/or face)
2. 2nd degree deep partial
3. area is from 1 to 10% BSA

All deep 2nd degree burn should be treated with the investigation product, Mepilex Ag/SSD (according to the randomization).

Exclusion Criteria:

* Burns "occurred" equal to or older than 36 hours
* Burns of chemical and electrical origin
* Clinically infected burn (as judged by the investigator)
* Subjects with lung injury or subjects being on a ventilator
* Treatment of the burn with an active agent before study entry. SSD is allowed up to 24 hours prior to randomization
* Subjects with dermatologic skin disorders or necrotizing processes
* Diagnosed underlying disease(s) (e.g. HIV/AIDS, cancer and severe anaemia) judged by the investigator to be a potential interference in the treatment
* Subjects with insulin dependent diabetes mellitus
* Subjects treated with systemic glucocorticosteroids, except Subjects taking occasional doses or doses less than 10mg prednisolon (day or equivalent
* Use of immunosuppressive agents, radiation or chemotherapy within the past 30 days
* Known allergy/hypersensitivity to any of the components (SSD , Ag glycerin, monostearate, glycerol, cetearyl alcohol, leveling agent O, albolene, light liquid paraffin, ethylparaben/ silicone, polyurethane foam pad containing a silver compound, activated carbon)of the investigation products
* Subjects with physical and/or mental conditions that are not expected to comply with the investigation
* Participation in other clinical investigation(s) within 1 month prior to start of the investigation
* Pregnancy (pregnancy test needed if they do not use contraceptive)
* Previously randomized to this investigation (PUMA 418

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zia Zhaofan, Principal Investigator — Changahai Hospital of Shanghai
Locations (9):
- China (9):
  - The 1st People's Hospital of Foshan, Guangdong, Guangdong
  - Guangzhou red Cross Hospital, Guangzhou, Guangdong
  - The First People's Hospital of ZhengZhou, Zhenzhou, Henan
  - The 3rd People's Hospital of Wuxi, Wuxi, Jiangsu
  - Beijing Jishuitan Hospital, Taiyuan, Shanxi
  - Xijing Hospital, XiAn, Shanxi
  - The 2nd affiliated Hospital of KunMing Medical college, Kunming, Yunnan
  - Beijing Children's Hospital, Beijing
  - Changhai Hoospital of Shanghai, Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- SSD Ag Cream: Silver Sulphadiazine Ag cream
  Silver sulphadiazine: Cream
Period: Overall Study
Arm/Group | Mepilex Ag | SSD Ag Cream
Started | 75 | 87
Completed | 66 | 74
Not Completed | 9 | 13
Not completed — Lost to Follow-up | 3 | 4
Not completed — Subject shedding | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Other | 4 | 4

BASELINE CHARACTERISTICS:
Population: ITT population/Safety population was chosen for the Overall Baseline Participants. ITT includes all Subjects, subject to at least one post-randomisation treatment and that provide some data for the primary endpoint.
Groups:
- Mepilex Ag: Mepilex Ag consists of a Safetac® soft silicone wound contact layer, a grey absorbent polyurethane foam pad containing a silver compound, activated carbon, and a vapour permeable waterproof film.
  Mepilex Ag: Dressing
- SSD Ag Cream: Silver Sulphadiazine Ag white cream, 1% SSD Ag, 40g/tube
  Silver sulphadiazine: Cream
- Total: Total of all reporting groups
Arm/Group | Mepilex Ag | SSD Ag Cream | Total
Number analyzed (Participants) | 71 | 82 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 6 | 9
  Between 18 and 65 years | 68 | 76 | 144
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (12.3) | 35.4 (13.2) | 36.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 25 | 41
  Male | 55 | 57 | 112
Region of Enrollment [Number; unit: participants]
  China | 71 | 82 | 153

OUTCOME MEASURES:

1. Primary Outcome: Time to Healing
Description: Healing will be defined as number of days
Time Frame: 4 weeks
Population: ITT population/Safety population. ITT includes all Subjects, subject to at least one post-randomisation treatment and that provide some data for the primary endpoint.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mepilex Ag | SSD Ag Cream
Number analyzed (Participants) | 71 | 82
days | 16 (7.27) | 17 (6.39)

2. Secondary Outcome: Percent of Burn Epithelised/Healed
Description: Healing will be defined as 95% or more epithelialisation
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of study burn healed
Arm/Group | Mepilex Ag | SSD Ag Cream
Number analyzed (Participants) | 71 | 82
percentage of study burn healed | 87.1 (29) | 85.2 (27.8)

3. Secondary Outcome: Number of Dressing Changes
Description: Number of dressing changes including first assembly
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: applications
Arm/Group | Mepilex Ag | SSD Ag Cream
Number analyzed (Participants) | 71 | 82
applications | 3.1 (1.86) | 14.0 (13.0)

4. Secondary Outcome: % of Study Burn Healed After One Week
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: percentage of study burn healed
Arm/Group | Mepilex Ag | SSD Ag Cream
Number analyzed (Participants) | 71 | 82
percentage of study burn healed | 44.3 (37.4) | 27.0 (30.7)

ADVERSE EVENTS:
Arm/Group | Mepilex Ag | SSD Ag Cream
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/82
Other Adverse Events (participants affected / at risk) | 0/71 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No